CLINICAL TRIAL: NCT01474356
Title: HDR Brachytherapy Combined With Interstitial Hyperthermia 500 kHz in Locally Advanced Cervical Cancer Patients. A Prospective Clinical Trial
Brief Title: Hyperthermia Combined Brachytherapy in CCU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTCCU01
Record Dates: First submitted 2011-10-20; First posted 2011-11-18 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Cervical Cancer
Keywords: brachytherapy; interstitial hyperthermia; cervical cancer; side effects; Locally advanced cervical cancer patients
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BT (brachytherapy) (No Intervention): Cervical cancer patients after the treatment with external beam radiotherapy combined with chemotherapy. In this group of patients, interstitial brachytherapy only was performed.
  Interventions: Other: hyperthermia
- BTHT (brachytherapy and hyperthermia) (Experimental): Cervical cancer patients after the treatment with external beam radiotherapy combined with chemotherapy. In this group of patients, interstitial brachytherapy with interstitial hyperthermia was performed.
  Interventions: Other: hyperthermia

INTERVENTIONS:
Other: hyperthermia — 45 minutes of interstitial heating 42.5-49°C during the interstitial brachytherapy

SUMMARY:
The aim of this randomised trial was to investigate whether hyperthermia (HT) combined with interstitial brachytherapy (ISBT) has any influence on local control (LC), disease-free survival (DFS), or acute and late side effects in patients with advanced cervical cancer. Vaginal symptoms were assessed by SOMA score, bladder and rectum symptoms by EORTC/RTOG score. Following the completion of radiochemotherapy, consecutive patients with cervical cancer (FIGO stage II - III) were randomly assigned to two treatment groups, either ISBT alone or ISBT combined with interstitial hyperthermia (ISHT). A total of 205 patients were included in the statistical analysis. Once a week, HT, at a temperature above 42.5°C, was administered for 45 minutes before and during the HDR BT. Follow-up examinations were scheduled at 6 weeks after the completion of BT, every 3 months during the first 2 years, and every 6 months throughout the next 3 years. If relapse was suspected, biopsies were obtained from these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with locally advanced cervical cancer FIGO stage II - III
* signed informed consent for participation in the study

Exclusion Criteria:

* patients with FIGO stage I and IV
* patients with poor performance status with contraindications for radical treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2006-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
LC | Follow up was scheduled every 3 months. Preliminary results after 3 years.
  When local relapse was suspected, biopsy was obtained.

SECONDARY OUTCOMES:
Late side effects | Follow up was scheduled every 3 months. Preliminary results after 3 years.
  EORTC\ERTOG scale for rectum and bladder and SOMA scale for vagina
Early complications of BT procedure | 24 hours after BT procedure
  Reporting the episodes of perforation and bleeding.
DFS | Follow up was scheduled every 3 months. Preliminary results after 3 years.
  CT, RTG, MRJ, SCC are performed to detect metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Żółciak-Siwińska, PhD, Study Chair — M. Sklodowska-Curie Memorial Cancer Centre and Institute, Roentgena 5, 02-781 Warsaw, Poland
Locations (1):
- Maria Skłodowska-Curie Memorial Cancer Center and Institute, Warsaw, Poland